CLINICAL TRIAL: NCT03959215
Title: Back in the Game: a Smartphone Application to Support Athletes Returning to Sport After Serious Injury
Acronym: BANG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Research Council for Sport Science (Other); American Orthopaedic Society for Sports Medicine (Other); Region Östergötland (Other); Psykologpartners (Unknown)
Responsible Party: Principal Investigator, Clare Ardern, Senior Researcher, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2019-0174
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Knee injuries; Anterior cruciate ligament injuries; Telemedicine
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care + Back in the Game (Experimental): Smartphone-delivered cognitive behavioural therapy to support confidence to return to sport + usual post-operative physiotherapy rehabilitation
  Interventions: Behavioral: Back in the Game
- Usual care (Active Comparator): Usual post-operative physiotherapy rehabilitation
  Interventions: Other: Usual rehabilitation care

INTERVENTIONS:
Behavioral: Back in the Game — A six-month programme of cognitive-behavioural therapy delivered by smartphone application. The intervention commences in the first week after ACL reconstruction. The smartphone app is delivered in parallel with usual rehabilitation care.
  Usual rehabilitation care: all participants will be referred to physiotherapy following ACL reconstruction. Overall treatment aims, content and progressions of rehabilitation will follow current clinical guidelines. The choice of specific therapies, exercises and the number of treatment sessions needed to achieve the treatment aims is at the clinical discretion of the treating physiotherapist.
  Arms: Usual care + Back in the Game
Other: Usual rehabilitation care — Following ACL reconstruction, as per routine clinical practice, all participants will be referred to physiotherapy. Overall treatment aims, content and progressions of rehabilitation will follow current clinical guidelines. The choice of specific therapies, exercises and the number of treatment sessions needed to achieve the required treatment aims is at the clinical discretion of the treating physiotherapist.
  Arms: Usual care

SUMMARY:
Returning to sport is one of the primary concerns of athletes following injury. Yet, after serious injury, up to 50% of athletes do not return to competitive sport. Psychological factors play an important role in the athlete's return to sport after anterior cruciate ligament (ACL) reconstruction, and physical and psychological readiness to return to sport often do not coincide. There are currently no easily accessible programs for non-professional athletes to help address the psychological factors that impact on their return to sport after injury.

The aim of this trial is to test whether a smartphone application (app) delivering cognitive-behavioural therapy to address psychological factors including fear, confidence and recovery expectations, is effective for improving the number of people who return sport following ACL reconstruction.

We hypothesise that patients who use the app in addition to receiving usual rehabilitation care after ACL reconstruction will return to sport in greater numbers than patients who receive usual rehabilitation care only.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary anterior cruciate ligament rupture
* Time between injury and anterior cruciate ligament reconstruction not greater than 12 months
* Playing contact pivoting or non-contact pivoting sport at least twice per week prior to anterior cruciate ligament injury
* Intend to return to sport following anterior cruciate ligament reconstruction
* Age 15 to 30 years at anterior cruciate ligament injury
* Normal/healthy contralateral knee

Exclusion Criteria:

* Collateral ligament injury requiring surgery
* Posterior cruciate ligament injury
* Meniscus injury/treatment that requires alteration to usual rehabilitation programme
* Articular cartilage injury/treatment that requires alteration to usual rehabilitation programme
* Previous anterior cruciate ligament injury to either knee
* Injury to either leg that required medical care during the previous 12 months
* Other injury or illness that could affect knee rehabilitation
* Taking medication for mental health problems

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Return to sport rate | At 1 year
  Rate of return to the preinjury sport and level of participation

SECONDARY OUTCOMES:
Self-reported participation in leisure time physical activity | Every two weeks to 1-year follow-up; every month from 1 to 2 years follow-up
  Every two weeks, participants will report the number of minutes spent in physical activity and the number of physical activity sessions including, but not limited to knee physiotherapy/rehabilitation sessions, active recreation, training and competitive sport.
New knee injuries | Every 2 weeks from 10 weeks to 1-year follow-up; every month from 1 to 2 years follow-up
  We will use an 'all complaints' definition of injury - participants self-report any new knee problems that have occurred during the surveillance window.
ACL- Return to sport after injury scale score | 3 months, 6 months, 9 months, 1 year, 2 years
  The ACL-Return to sport after injury scale (ACL-RSI) is a 12-item scale designed to measure psychological readiness to return to sport after ACL injury. Scores range from 0 to 100; higher scores indicate greater psychological readiness to return to sport.
Knee Self-Efficacy Scale 'future' domain | Before surgery, 1 year, 2 years
  The 'future' domain of the knee self-efficacy scale comprises 4 questions to assess self-efficacy related to future knee function:
  1. How certain are you that you can return to the same physical activity level as before the injury?
  2. How certain are you that you would not suffer any new injuries to your knee?
  3. How certain are you that your knee would not 'break'?
  4. How certain are you that your knee will not get worse than before surgery?
  Each question is scored on a 0-10 scale (higher scores represent greater self-efficacy). The domain score is the mean of responses to the four questions.
Motivation to participate in leisure time physical activity | 3 months, 6 months, 9 months
  We will use three questions all measured on a 1-10 scale, where higher scores represent higher motivation:
  1. How important is it for you to return to the same sport or recreation activity as before your knee injury?
  2. Do you think it is possible for you to return to the same sport or recreation activity as before your knee injury?
  3. How much time and effort are you willing to invest to return to the same sport or recreation activity as before your knee injury?
ACL-Quality of Life scale score | 1 year, 2 years
  The ACL-QoL is a 30-item scale to measure knee-related quality of life following ACL injury. Scores range from 0 to 100; higher scores indicate greater knee-related quality of life.
Self-reported knee function (Single Assessment Numeric Evaluation (SANE) and International Knee Documentation Committee (IKDC) subjective knee form) | Before surgery, 6 months, 1 year, 2 years
  The item wording for SANE is: "on a scale from 0-100, where 100 represents the best, how would you rate your knee today?" The IKDC subjective knee form is a 19-item condition-specific measure. The IKDC is scored out of 100 points, with a higher score indicating superior self-reported knee function.
Thigh muscle strength | 1 year
  We will use an isokinetic dynamometer to measure quadriceps and hamstrings concentric and eccentric peak torque.
Hopping performance | 1 year
  We will measure the single hop for distance, triple hop for distance and side hop test for the affected and unaffected sides. The single hop for distance is the maximum distance the person can hop from a stationary starting position. The triple hop for distance is the maximum distance the person can hop with three successive hops from a stationary starting position. The side hop test is the number of hops the person can complete side-to-side over a 40cm strip of tape, in a 30 second period. If the person steps on the tape, the test must stop and be repeated.
Adherence to physiotherapy | Every 2 weeks that the person is completing rehabilitation
  Participants will self-report the number of supervised physiotherapy sessions, number of home-based exercise sessions and the number of gym-based exercise sessions completed in the previous 2 weeks.
Adherence to smartphone intervention | At 6 months
  We will count page views for different types of content (including Vimeo for video content, Soundcloud for audio content).
Hospital Anxiety and Depression Scale score | Before surgery
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale that measures psychological distress. Scores range from 0 to 21; higher scores indicate greater psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Clare L Ardern, PhD, Principal Investigator — Department of Family Practice, University of British Columbia
Locations (7):
- Sweden (7):
  - Eksjö Hospital, Eksjö
  - Capio Lundby, Gothenburg
  - County Hospital Ryhov, Jönköping
  - Linköping University Hospital, Linköping
  - Capio Artro Clinic, Stockholm
  - Praktikertjänst Orthopaedics, Stockholm
  - Värnamo Hospital, Värnamo

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for the primary and secondary outcomes will be shared with researchers whose proposed use has been approved by an independent review committee, for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Data must be requested through the Swedish National Data Service. Data will be available within 6 months of study completion and are available indefinitely.
Access Criteria: Requestors will be required to sign a Data Access Agreement.
URL: http://snd.gu.se

REFERENCES:
- [Background] Ardern CL, Kvist J; BANG Trial Group. BAck iN the Game (BANG) - a smartphone application to help athletes return to sport following anterior cruciate ligament reconstruction: protocol for a multi-centre, randomised controlled trial. BMC Musculoskelet Disord. 2020 Aug 8;21(1):523. doi: 10.1186/s12891-020-03508-7. PMID 32770983
- [Background] Ardern CL, Hooper N, O'Halloran P, Webster KE, Kvist J. A Psychological Support Intervention to Help Injured Athletes "Get Back in the Game": Design and Development Study. JMIR Form Res. 2022 Aug 9;6(8):e28851. doi: 10.2196/28851. PMID 35943769
- [Derived] Ringberg M, Eldh AC, Ardern CL, Kvist J. Athletes' experiences of using a self-directed psychological support, the BAck iN the Game (BANG) smartphone application, during rehabilitation for return to sports following anterior cruciate ligament reconstruction. BMC Sports Sci Med Rehabil. 2023 Sep 19;15(1):113. doi: 10.1186/s13102-023-00731-2. PMID 37726848

DOCUMENTS (1):
  • Informed Consent Form (2020-04-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT03959215/ICF_000.pdf